CLINICAL TRIAL: NCT01308775
Title: A Pilot Study Comparing a Patient-Centered Symptom Reporting Follow Up Program (SIS.NET) to Standard Care in Patients Who Have Completed the Acute Phase of Treatment for Early Breast Cancer
Brief Title: Comparing (SIS.NET) to Standard Care in Patients Who Have Completed the Acute Phase of Treatment for Early Breast Cancer
Acronym: CC077515
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CC077515
Record Dates: First submitted 2011-02-24; First posted 2011-03-04 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Breast Cancer
Keywords: SIS.NET
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SIS.NET, Routine Follow up (Active Comparator)
  Interventions: Behavioral: SIS.NET, Routine Follow-up

INTERVENTIONS:
Behavioral: SIS.NET, Routine Follow-up — * SIS.NET - One or two oncology related clinic visits per year (as recommended by the American Society of Clinical Oncology breast cancer follow up guidelines (18)), with additional access to oncology care driven by ongoing review of patient's self reported symptoms through web-based questionnaires.
  * Routine follow up care with appointment frequency determined by the treating medical oncologist or oncology/breast surgeon. Patients complete the same web-based symptom questionnaires within 30 days of a scheduled clinic visit but the results are not reviewed until their clinic visit.

SUMMARY:
This is a pilot study that will compare two systems of breast cancer follow up care and will evaluate a number of parameters indicating quality and efficiency of care delivery as well as patient satisfaction with care. Approximately 100 breast cancer patients who have completed the acute phase of treatment will be randomized to one of two follow up care plans.

DETAILED DESCRIPTION:
Over 200,000 women were diagnosed with breast cancer in the year 2006. Many of these women will be rendered free of cancer, but will need ongoing disease specific care and surveillance. The estimated number of breast cancer survivors in the year 2003 was 2.3 million (1). With outcomes improving after the diagnosis of early breast cancer, the number of breast cancer survivors in follow up care will continue to increase and eventually result in an unmanageable load on the subspecialties of medical and surgical oncology. Most of these patients continue to be seen by an oncology specialist for at least five years after their cancer diagnosis, but this type of follow up may not be necessary or optimally utilized.

Alternate Strategies for Health Care Delivery Studies suggest that oncology follow up care is costly to the health care system no matter who the provider is, and in some cases, diagnostic tests are overused (2). In a randomized trial of 296 women with a history of breast cancer in Great Britain, transfer of routine follow-up care to a family physician did not result in an increase in the time to diagnosis of recurrence (3). Patient satisfaction was greater and health service costs were less, and anxiety and health related quality of life were unaffected (4, 5). A similar multicenter trial of 968 early-stage breast cancer patients in Canada who had completed adjuvant treatment randomized patients to follow up in a cancer center or with their own family physician (6). This study found no statistically significant differences in number of recurrences, deaths, recurrence related serious clinical events, or patient reported health-related quality of life questionnaires between the groups. While transferring oncology follow-up care back to primary care physicians seems a reasonable alternative, the shortage of primary care physicians in certain regions of the US and around the world, limits this approach (7, 8). A study in Sweden compared nurse-led follow-up vs. physician follow-up in 264 consecutively selected women with newly diagnosed Stage I or II breast cancer (9). Outcomes included measures of patient well-being, satisfaction, access to medical care, and medical safety. Questionnaires containing the Hospital Anxiety and Depression Scale (HADS), and the Satisfaction and Accessibility (SaaC) scale were obtained at baseline and twice a year over a period of 5 years. Number of contacts with health care services, number of diagnostic procedures, and time to recurrence or death were monitored. Ratings of HADS and SaaC scales did not show any statistically significant differences between the follow-up groups. The levels of anxiety and depression were generally low, and levels of patient satisfaction high. There were no differences between the groups concerning time to recurrence or death suggesting that follow-up care with an experienced nurse professional is safe and effective.

Various strategies have been studied to evaluate alternatives to routine clinic visits and referrals to subspecialists in order to improve access to care and to lower health care costs. One such study tested the hypotheses that virtual outreach would reduce number of contacts with the health care system, reduce the number of medical tests and interventions, and have a positive impact on patient satisfaction. A randomized controlled trial was conducted which compared standard outpatient referral to joint teleconsultations between general practitioners (GP), specialists, and patients (10). Patients randomized to virtual outreach underwent a joint teleconsultation, in which they and their GP consulted with a hospital specialist via a videolink. In this study, patients in the virtual outreach group were more likely to be scheduled for a follow-up appointment, but fewer tests and investigations were ordered. In the 6-month period following the initial consultation, there were no significant differences in number of contacts or outpatient visits with GP, inpatient stays, procedures, or prescriptions between the randomized groups. Patient satisfaction was greater after a virtual outreach consultation, and patient enablement and the physical and psychological scores of the Short Form-12, did not differ between the randomized groups. Interestingly, health care costs over 6 months were greater for the virtual outreach consultations than for conventional outpatients, but overall cost, time, and productivity savings to patients were identified. This study represents an example of how technology can be utilized to streamline care and provide more patient centered services, but that these services may not save money overall in the health care system. The need to assess the cost-effectiveness and patient outcomes of alternate surveillance and follow up strategies was recently highlighted in a review article by Tolaney (11).

UCSF and Dynamic Clinical Systems (DCS) Collaboration The UCSF Breast Care Center has embarked upon collaboration with Dynamic Clinic Systems to implement a computer based, patient centered system of symptom reporting and data collection to improve clinical care to our patients and generate databases of patient reported symptoms and outcomes information for research purposes. Dynamic Clinical Systems (DCS) is a provider of real-time Web-based applications focusing on the patient-clinician interaction. The DCS approach enables patients to provide health data electronically. Clinicians may use this data for research, medical documentation, and registries depending on the type of data collected and the consent of the patient.

Through this system, patients will report their own health information via the DCS web-based Integrated Survey System (ISS). The process is as follows: A real-time interface downloads appointments from the hospital scheduling system into ISS. Survey groups are automatically scheduled based on pre-defined timing parameters. Prior to sending the patient their first survey, each patient will be called and welcomed to the program and asked if they use the internet. If they do, they will be given instructions for completion of surveys at home. If they need assistance, they will be given an appointment to come to our resource center and work with our staff member to complete the survey. The patient will be notified (via automatically-generated email from ISS or hospital letter/phone) to either sign on and take the survey from home or come to clinic early to take the survey. Once logged in, the patient has the opportunity to indicate online consent (to be approved by CHR) to share data for research purposes. An analyst will monitor the progress of survey completion and will call any patient whose surveys are not complete prior to their clinic appointment to facilitate survey completion. At the end of the process, a patient summary report is generated in ISS displaying a summary of patient survey answers, longitudinal comparisons of previous surveys, red flags and warnings, and quality measures. The clinician uses this report during the clinic visit to focus the discussion on highlighted items.

DCS is a service vendor who has built and who services the online-questionnaire platform. All content in the questionnaires has been created and reviewed by the investigators at UCSF (with the exception of standardized surveys such as the SF-36 and other validated questionnaires). Other than this, the DCS has no role in this study, and it does not receive or have access to information regarding study outcomes (such as in terms of patient visits or interventions) from either arm of the study.

We plan to implement and evaluate a comprehensive survivorship program, supported by this interactive web-based system for reporting physical and psychological symptoms. The system will capture structured data that then can be used to drive translation of research findings to improve care for survivors. The System for Individualized survivorship care, based on patient Self-reported data, with review by Nurse practitioners, targeted Education, and Triage to appropriate services to improve symptom management and outcomes will be called SIS.NET

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with Stage I to Stage III breast cancer that have completed their acute phase of treatment. (This includes surgery, radiation, chemotherapy, or any experimental therapies offered in a clinical trial as adjuvant treatment.)

   * Patients who received chemotherapy must be 6 months out from completion of chemotherapy.
   * For patients who receive adjuvant hormonal therapy (with or without prior chemotherapy), patients must be 3 months out from initiation of hormonal therapy.
   * For patients who do not receive adjuvant chemotherapy or hormonal therapy, patients must be 3 months out from surgery and radiation therapy.
2. Patients must have recovered from all serious side effects of acute phase of treatment for breast cancer.
3. Patients must be willing to complete symptom reporting questionnaires at the intervals assigned by their care group.
4. Patients must have hematologic, cardiac, hepatic, and renal function that are back to their pre-treatment values.
5. Patient must be able to read and speak English sufficiently to complete symptom reporting questionnaires and discuss details of symptoms and health status over the telephone.
6. Patient must have access to a computer on which to complete the on-line surveys or must be willing to come to the UCSF Cancer Resource Center to complete questionnaires at the intervals assigned by their care group.

Exclusion Criteria:

1. History of severe depression or an anxiety disorder that is felt to interfere with a patient's ability to accurately self-report symptoms.
2. Complications from breast surgery or reconstruction, or from chemotherapy or radiation that may require regular ongoing clinic visits for physical and/or laboratory evaluation.

   -

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2011-01; Primary Completion 2014-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the time to evaluation of breast cancer or breast cancer treatment-related symptoms, between patients enrolled in a system of symptom-based, patient centered follow-up care (SIS.NET) and patients receiving standard follow up care | 18 months
  This aim will determine which follow up care system provides more timely assessment and management of patient reported symptoms. Currently, patients may wait up to 2 weeks or more to be seen in clinic if they experience a new symptom in between regularly scheduled appointments. Our goal is to assess a patient's newly reported symptom in 3 business days or less.

SECONDARY OUTCOMES:
To compare the number of oncology and primary care provider clinic visits, other subspecialty clinic visits, emergency room visits and phone calls to oncology related health care providers and triage nurses. | 18 months
  To compare the number of oncology and primary care provider clinic visits, other subspecialty clinic visits, emergency room visits, and phone calls to oncology related health care providers and triage nurses between patients in SIS.NET vs. standard follow-up care.
To compare the number of breast cancer and breast cancer treatment related diagnostic tests between patients enrolled in a computerized system and patients receiving standard follow up care. | 18 months
  To compare the number of breast cancer or breast cancer treatment related diagnostic tests. Current ASCO follow up guidelines do not recommend the use of routine laboratory tests, tumor markers, or radiologic examinations (other than annual mammograms) for breast cancer follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Melisko, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States

REFERENCES:
- [Derived] Wheelock AE, Bock MA, Martin EL, Hwang J, Ernest ML, Rugo HS, Esserman LJ, Melisko ME. SIS.NET: a randomized controlled trial evaluating a web-based system for symptom management after treatment of breast cancer. Cancer. 2015 Mar 15;121(6):893-9. doi: 10.1002/cncr.29088. Epub 2014 Dec 2. PMID 25469673